CLINICAL TRIAL: NCT05402358
Title: Acceptability and Feasibility of Groups for Specific Versus Mixed-diagnosis Patients of Long-term Conditions
Brief Title: Groups for Specific vs Mixed Diagnosis Patients of Chronic Conditions
Status: Completed | Type: Observational
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Holly Martin-Smith, Postgraduate Research Student, University of Stirling
Other Study IDs: 274421
Record Dates: First submitted 2022-02-07; First posted 2022-06-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Diabetes; Cardiovascular Diseases; Skin Diseases; Rheumatic Diseases; Mental Health Issue
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Skin Diseases; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Specific-Diagnosis: There were four specific-diagnosis groups covering four specialities: Dermatology, Rheumatology, Diabetes and Cardiology. Participants were categorised into these groups dependent on the speciality from which the referral originated or the participants primary condition. Participants attending a specific-diagnosis group were required to have a diagnosis relating to that speciality. All participants received the Living Well with a Long-Term Condition intervention
  Interventions: Other: Acceptance and Commitment Therapy Group Intervention
- Mixed-Diagnosis: There were four mixed-diagnosis groups; participants who do not fall into the above specialities, or had number of co-morbid conditions, or were unable to attend the specified dates for any of the four specific-diagnosis groups, were invited to attend a mixed-diagnosis group.All participants received the Living Well with a Long-Term Condition intervention
  Interventions: Other: Acceptance and Commitment Therapy Group Intervention

INTERVENTIONS:
Other: Acceptance and Commitment Therapy Group Intervention — The intervention consists of 7, 2-hour weekly sessions. Session 1 focused on introductions, outlining sessions and sharing experiences. Session 2 introduced key techniques used in the psychological approach (ACT) including mindfulness and understanding difficult thoughts and feelings. Session 3 explored ideas of primary and secondary suffering and reviewed the workability of current coping strategies. Session 4 asked participants to clarify their own personal values. Session 5 focused on goal setting and utilising problem solving skills. Session 6 considered barriers to change including assertiveness communication skills. Session 7 reviewed topics covered over the 6 weeks previously and explored pacing and preparing for setbacks. Finally a follow up 8 weeks later brought participants back for a reunion to review progress with goals and offer an opportunity to address any ongoing issues.

SUMMARY:
Does a group programme already delivered in routine practice to patients who share a diagnosis from the same medical speciality (i.e. specific-diagnosis) show equal effectiveness when modified for patients with diagnoses from a range of medical specialities (i.e. mixed-diagnosis)?

A large number of people live with a long-term condition (LTC) and the burden of living with a LTC is recognised on a societal and individual level. Links between LTCs and poorer mental health increase demand on psychological services. Consequently new initiatives try to reduce waiting times and increase the capacity of these services. Group programmes use resources efficiently and have been applied across a range of medical specialities. A clinical health psychology service has adopted a group programme based on a well evidenced psychological therapeutic approach called Acceptance and Commitment Therapy (ACT), for patients with dermatology conditions showing promising outcomes. However, the investigators want to compare whether similar outcomes can be achieved with patients from a range of specialities.

The investigators conducted quantitative and qualitative research to answer the research questions a) Does an Acceptance and Commitment Therapy group intervention for specific-diagnosis groups suggest similar effectiveness in health-related quality of life, illness beliefs and psychological distress versus mixed-diagnosis groups? b) Is there a difference in feasibility and acceptability of an Acceptance and Commitment Therapy intervention between specific-diagnosis groups versus mixed-diagnosis groups? c) What are health professionals' views on the acceptability and feasibility of specific-diagnosis versus mixed-diagnosis groups and their experiences of working with patients who have attended such groups?

Participants were recruited from the Clinical Health Psychology waiting list at a UK NHS Trust. Participants attended 7, two-hour weekly sessions and an 8 week follow-up 'reunion', and completed health related quality of life, illness perceptions, depression and anxiety questionnaires pre and post intervention. Patient participants and health professional participants (facilitators and referrers) were invited to attend focus groups to discuss their views and experiences.

DETAILED DESCRIPTION:
Design

A mixed methods pilot and feasibility study was selected and applied. Mixed methods were selected as it integrates rich and comprehensive data from a quantitative and qualitative approach, to answer the overall studies research questions:

1. Is there a difference in feasibility and acceptability of an online ACT intervention between specific-diagnosis versus mixed-diagnosis groups?
2. What are health professionals' views on the acceptability and feasibility of specific-diagnosis versus mixed-diagnosis groups and their experiences of working with patients who have attended such groups?
3. Do the results of this small pilot and feasibility study suggest similar effectiveness in health-related quality of life, illness beliefs and psychological distress in specific-diagnosis versus mixed-diagnosis groups? We delivered online groups. Quantitative data collected from attendance records, and qualitative data collected from qualitative interviews with participants who took part in the intervention, addressed research question 1. Qualitative data collected from qualitative interviews with health professionals who facilitated the intervention, and health professionals who referred patients to the intervention, addressed research question 2. Finally, quantitative data collected from psychometric measures, addressed the third research question.

Study participants

Patient participants were recruited from the Clinical Health Psychology GM team waiting list, or by being made aware of the groups by health professionals working within specialities covered by the GM team. As per routine clinical practice, patients on the waiting list were invited to attend the group intervention via letter or during a routine waiting list check-in review. The waiting list was regularly reviewed so for each scheduled group, only new appropriate patients on the waiting list were sent invites (i.e., each patient only received one invite to respect their choice not to participate).

We had planned for potential patient participants to be able to self-refer to the clinical team. Self-referrals were expected from patients who saw an advertising poster placed in the waiting rooms of the hospital specialties the GM team covered. Since face-to-face healthcare was extremely limited during the recruitment period, posters were not used.

All interested participants received a telephone screening consultation, including a brief psychological assessment, to check each participant was suitable and that they met inclusion criteria. This assessment informed patients about the research study in line with details provided in the participant information sheet.

If after this telephone screening assessment with a clinical team member a participant met the inclusion criteria, and wished to continue, they were allocated to the intervention and invited into one of the group conditions, dependent on their diagnosis. Written consent was obtained at the start of the intervention.

The group intervention was still offered to any patient who did not want to take part in the research. If a patient was not suitable, they were offered appropriate alternative treatment as deemed necessary by the assessing clinician.

At the last session of the intervention, patient participants recruited to the research were invited via email to take part in a qualitative interview to explore their views and experiences.

Two types of health professional participants were recruited:

(A) Those who facilitated/delivered the intervention (B) Those who referred patients to the intervention Facilitators were invited via email to take part in an online focus group, and referrers were invited via email to take part in online individual interviews. These explored health professional participants views of the intervention and experiences of working with patients in relation to the groups. The only facilitator who was excluded from participating was the main researcher due to potential researcher bias. All health professional participants were informed about the research study and given a participant information sheet, prior to consenting to take part.

Procedure

The online ACT group intervention was delivered to two group conditions, specific-diagnosis and mixed-diagnosis. Each group condition had four intervention group programmes, totaling eight groups overall. Prior to the COVID-19 pandemic it was standard practice to deliver groups face-to-face, however, government enforced restrictions meant that this was not allowed particularly during national lockdowns. Hence the delivery format was changed to online.

The ACT group intervention was called 'Living Well with a Long-Term Condition' and was adapted from the Brassington et al., (2016) 'Better Living with Illness' protocol. A clinician handbook, and participant workbook , was developed that could be used for both group conditions. These materials were adapted by the researcher and other members of the GM team, all of whom had received specialist training in ACT. Each group was delivered online using a platform called 'Microsoft Teams'. The intervention was facilitated by two qualified clinicians. The intervention consisted of 8, 2-hour sessions. Sessions 1-7 were delivered on a weekly basis, followed by a gap of 8 weeks, before the final 'reunion' session. In summary the sessions covered the six core processes of ACT, included experiential exercises, and allowed for group discussions to share experiences and learning between participants.

Online 'screen share' materials were developed so that facilitators could guide participants through the session content. Microsoft teams had features that were utilised to support the group sessions such as camera, mute, raise hand, text chat and share screen functions. Participants were encouraged to have their camera on during group sessions, but it was not mandatory (to respect privacy and confidentiality). At the end of the sessions, facilitators remained logged into the meeting for 15 minutes, to allow for any participants to answer questions privately. Telephone calls were also offered, should any participants have any questions which could be requested via email. Summary emails were sent following each session which included links to access any exercises as part of their home-practice between sessions.

Participants who missed sessions were signposted to read through information provided in their participant workbook and offered a telephone consultation to talk through any missed content. It was decided that if anyone missed the first two sessions consecutively, they were transferred to the next mixed-diagnosis group available or returned to the waiting list. This decision was based on the potential to cause disruption to the group dynamics, whereby social relationships would likely have already been established, making it difficult for a new person to interact with the group and feel part of the 'group spirit', which may also negatively impact a patient's own wellbeing. Unfortunately, resources did not allow multiple specific-diagnosis groups to run hence the option to transfer to another specific-diagnosis group was not possible.

Measures

Psychometric questionnaires were completed by patient participants to assess psychological distress, illness perceptions and health-related quality of life at three different timepoints, baseline (pre-treatment), session 7 (post-treatment) and session 8 (8-week follow-up).

Other quantitative measures to assess the feasibility and acceptability of the intervention to the patient participants included eligibility, recruitment, retention, true completion, and intervention adherence rates.

We collected qualitative data with patient participants and health professional participants.

Patient qualitative interviews

Patient participants who had consented to take part in the research were invited via email to take part in online focus groups and individual interviews using microsoft teams. These were moderated by a research assistant who had an honorary contract as a volunteer assistant psychologist with the Clinical Health Psychology service. The research assistant was provided with training on how to conduct focus groups and individual interviews, and was supervised by the main researcher, who had prior qualitative research experience. Originally four focus groups were planned, two for each of the group conditions. To improve recruitment an amendment to the ethics was approved (20/NW/0125/AM01), to include individual interviews as well as focus groups to collect qualitative data from any participants who had been unable to take part in focus groups. Both interviews and focus groups are an evidenced based method of data collection for qualitative studies (Harrell & Bradley, 2009), the pros and cons for both were considered, and it was concluded that this additional alternative method of data collection allowed for greater flexibility to arrange interviews at times to suit all participants busy schedules.

Participants were invited via email by the researcher and were given a participant information sheet. Those who took part provided written consent. All qualitative interviews were audio-recorded, focus groups lasted no longer than 2 hours and individual interviews lasted no longer than 30 minutes. A topic guide was used to elicit participants views and experiences of taking part in the intervention, as well as thoughts on the intervention being delivered to the two group conditions.

Health professional interview

One focus group was conducted with the facilitators of the intervention. Individual interviews were conducted with the referrers. All qualitative interviews were held online using microsoft teams and moderated by the same research assistant as above. All health professionals were invited via email and given participant information sheets explaining that the focus group would last no longer than one hour and individual interviews no longer than 30 minutes. Two topic guides were developed, to gather the views and experiences of health professionals including their thoughts on the two group conditions. All health professionals who agreed to take part provided written consent and all qualitative interviews were audio-recorded.

Quantitative data

A mixed 2 by 3 ANOVA analysis was used, to compare the mean differences between groups on the outcome measures. These were split on a between subjects' factors (group condition), and a within subjects' factor (time, with three timepoints; T1-baseline, T2-post treatment and T3-8 weeks follow-up), with data assessed for homogeneity, normality and sphericity, and appropriate adjustments made when assumptions were violated.

Descriptive statistics reported eligibility, recruitment, retention, true completion, and intervention adherence rates.

Qualitative data

Qualitative data was analysed aligned to a deductive and inductive, reflexive thematic analysis approach (Braun & Clarke, 2006; 2019, 2020). This commonly used hybrid approach was deemed appropriate, to best meet the aims of the study and answer research questions. Initially a theory-driven concept, the TFA , was applied for the process of deductive thematic analysis. Following this an inductive approach allowed the development of themes from the data and allowed for a broader understanding of the data. It is acknowledged that the coding approach was collaborative (as it involved multiple researchers) and reflexive whereby researchers' 'read' the data based on personal theoretical assumptions, analytic resources and skill. Thus, interpretations reflect those of the researchers' own experiences, beliefs and biases which will have affected the development and generation of themes and inferences.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants needed to have a diagnosis of:

  1. A long-term condition relating to one of the four specific-diagnosis specialities (Dermatology, Rheumatology, Diabetes, or Cardiology) for the specific-diagnosis group.
  2. A long-term condition (from any of the hospital specialities that the General Medicine team covered) for the mixed-diagnosis group (including any of the specific-diagnosis specialities; dermatology, rheumatology, diabetes or cardiology).

Patient participants were also required to be 18 or over, English speaking and able to give informed consent to participate.

Exclusion Criteria:

* they were actively engaged with another psychological therapy or receiving active input from a secondary mental health service
* they had significant substance abuse difficulties
* they had severe and/or chronic mental health problem such as personality disorder where the interpersonal difficulties themselves are the required focus of an intervention
* they had a learning disability, at such a level that specialist skills would be required to deliver an intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9) | Baseline, week 8 and 8 week follow up
  Self-report measure of depression. Minimum value 0 to maximum value 27, a higher score indicating a worse outcome.
The General Anxiety Disorder Scale (GAD-7) | Baseline, week 8 and 8 week follow up
  Self-report measure of anxiety. Minimum value 0 to maximum value 21, a higher score indicating a worse outcome.
The Brief Illness Perception Questionnaire (BIPQ) | Baseline, week 8 and 8 week follow up
  Self-reported perceptions of health. Overall score is computed and higher scores indicate more negative perceptions of illness.
The RAND 36-item Health Survey 1.0 | Baseline, week 8 and 8 week follow up
  Self-reported health-related quality of life assessing eight domains. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Group attendance | Through intervention completion, for 8 sessions
  The numbers of participants recruited and retained (we will record attendance levels at group sessions)
Focus group and individual interviews with patient participants | After intervention completion, on average 12 weeks
  Explored the thoughts and feelings of participants from each group on what worked well and could be improved about all aspects of the intervention including a) the attractiveness, accessibility and acceptability of the intervention b) the group environment and ideas of being in a specific-diagnosis versus mixed-diagnosis group
Focus group and individual interviews with health professional participants | After intervention completion, on average 12 weeks
  Qualitative measure explored the thoughts and feelings of health professionals on specific-diagnosis and mixed-diagnosis groups and include the believed advantages and disadvantages and any changes noticed in patients that they have referred or worked with who complete the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Martin-Smith, Principal Investigator — University of Stirling
Locations (1):
- Salford Royal NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No